CLINICAL TRIAL: NCT05092867
Title: Reliability and Validity of a New Postoperative Track Assessment Tool - a Prospective Observational Study
Brief Title: Reliability and Validity of a New Postoperative Track Assessment Tool
Acronym: POTraTool
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Laurelie Perret, principal investigator, University Hospital, Geneva
Other Study IDs: 14032019
Record Dates: First submitted 2021-09-21; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Perioperative Complication
Keywords: Post-Anesthesia Care Unit; Intermediate Care Unit; Clinical pathways; Decision making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Po Tra tool — Healthcare workers filled the 2 VAS of the tool but it did not impact or change the care of the patient. (observational)

SUMMARY:
This prospective observational study investigated the validity and reliability of a new postoperative track assessment tool. We hypothesized, first, that this tool estimates the indication and benefit of a management in an intermediate care unit (IMC). Second, we hypothesized that a) health care providers of IMC or postoperative anaesthesia care unit (PACU) have similar estimations using this tool and b) that this estimation is accurately established in the first 2 hours.

DETAILED DESCRIPTION:
The tool includes 2 visual analog scale (VAS) scores estimating indication of an IMC admission and benefit of an IMC stay. The tool was tested in a PACU and in an IMC unit of a Swiss tertiary centre in 2019/2020 (before COVID pandemic). Three raters: one nurse, one physician in charge and the consultant physician, were asked to fill the VAS at the same time for each included patient. The score was done in the 2 first hours following admission in the unit and during the multi professional morning round at day 1.

Reliability was estimated by testing internal consistency (homogeneity), interrater reliability and agreement and test-retest validity (stability). Validity included content validity, construct validity and criterion validity.

ELIGIBILITY:
Inclusion Criteria:

* PACU patients admitted on Mondays
* IMC patients admitted 7:30am-7:30pm on weekdays

Exclusion Criteria:

* night admission
* PACU patient ASA < 3 or minor intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was a random sample from the PACU and IMC patients' population. Included patients' variables for demographic description of the population of interest and for the validity testing were: Age in years, gender (male / female), ASA physical score classification (ASA PS), do not resuscitate order (DNR), duration of intervention (min), severity of intervention (minor/intermediate/major), type of surgery (abdominal, orthopedic, trauma and other surgical and non-surgical interventions), elective or non-elective, palliative intervention, SAPS II (admission (2 h after arrival in IMC)), NEMS (admission (2 h after arrival) and during stay in IMC), SAS.
  Participating raters were voluntary health care providers working in the peri-interventional unit (PACU and IMC).
Sampling Method: Non-Probability Sample
Enrollment: 879 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Intermediate Care (IMC) indication (VASi) | 2019/2020
  Health care raters graded the IMC indication (or allocative efficiency) for each patient on a visual analog scale grading from 0 (very low indication of an IMC management) to 100 (very high indication of an IMC management), namely VASi.
Intermediate Care benefit (VASb) | 2019/2020
  Health care raters graded the IMC benefit (or health gain) for each patient on a visual analog scale grading from 0 (very low benefit from an IMC management) to 100 (very high benefit from an IMC management), namely VASb.

CONTACTS AND LOCATIONS:
Overall Officials: Walder, Professor, Study Director — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Perret L, Buclin CP, Courvoisier DS, Walder B. Reliability and validity of a new postoperative track assessment tool (PoTra-tool) as a decision-making aid: A prospective observational study. Eur J Anaesthesiol Intensive Care. 2025 May 29;4(4):e0076. doi: 10.1097/EA9.0000000000000076. eCollection 2025 Aug. PMID 40756574